CLINICAL TRIAL: NCT04232514
Title: A Open-label, Single Center Drug Interaction Study Between HEC74647PA Capsule and HEC110114 in Healthy Subjects
Brief Title: Drug-drug Interaction Study Between HEC74647PA Capsule and HEC110114 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEC74647-P-03
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Subjects will receive HEC74647 on Day 1~7 and Day13~19, co-administration with HEC110114 on Day13~19.
  Interventions: Drug: HEC74647; Drug: HEC110114
- Part B (Experimental): Subjects will receive HEC110114 on Day 1~7 and Day13~19, co-administration with HEC74647 on Day13~19.
  Interventions: Drug: HEC74647; Drug: HEC110114

INTERVENTIONS:
Drug: HEC74647 — Administered HEC74647 200 mg orally once daily in fed state
Drug: HEC110114 — Administered HEC110114 800 mg orally once daily in fed state

SUMMARY:
The purpose of this study is to evaluate the drug-drug-interaction (DDI), pharmacokinetics (PK) and tolerability of HEC74647 combined with HEC110114 in healthy subjects

DETAILED DESCRIPTION:
This is a 2-part study with each part is an open-label study in healthy adult subjects.

Total 28 subjects will be enrolled into the study and divided into 2 part (Part A and Part B), 14 subjects in each part. With each part, the subject will be receive study drug per the defined treatment periods of Day 1~7 and Day 13~19.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form before the trial and fully understand the contents of the trial, the process and possible adverse reactions.
* Be able to complete the study according to the trail protocol.
* Subjects (including partners) have no pregnancy plan within 3 months after the last dose of study drug and voluntarily take effective contraceptive measures.
* Male subjects and must be 18 to 45 years of age inclusive.
* Body weight ≥ 50 kg and body mass index（BMI）between 18 and 28 kg / m2, inclusive.
* Physical examination and vital signs without clinically significant abnormalities.

Exclusion Criteria:

* Use of >5 cigarettes per day during the past 3 months.
* Known history of allergy to study drugs，or allergies constitution ( multiple drug and food allergies).
* History of alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits or 100 mL of wine).
* Donation or loss of blood over 450 mL within 3 months prior to screening.
* 12-lead ECG with clinically significant.
* Positive for Viral hepatitis (including hepatitis B and C), HIV and syphilis.
* Subjects deemed unsuitable by the investigator for any other reason.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-22 (Actual)

PRIMARY OUTCOMES:
Adverse Events | From Days 1-26
  Incidence of adverse events
Cmax | Day 7-12 and Day 19-26
  Maximum plasma concentration of study drugs
AUC | Day 7-12 and Day 19-26
  Maximum plasma concentration of study drugs

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China